CLINICAL TRIAL: NCT02782429
Title: The Role of Ketamine in Preventing Cognitive Dysfunctions in Postoperative Period of Cardiac Surgery
Acronym: KeCoDy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Flavia orange (Other)
Collaborators: Rebeca Gonelli Albanez da Cunha Andrade (Unknown)
Responsible Party: Sponsor-Investigator, Flavia orange, Prof, Dr, Instituto Materno Infantil Prof. Fernando Figueira
Organization: Instituto Materno Infantil Prof. Fernando Figueira (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: IMIP
Record Dates: First submitted 2016-05-19; First posted 2016-05-25 (Estimated); Last update posted 2016-05-25 (Estimated); Status verified 2016-05

CONDITIONS: Delirium; Inflammation; Cognitive Disorders; Amnestic; Dementia
Keywords: ketamine; Cardiac Surgery; Neurocognitive Disorders
MeSH Terms: conditions — Delirium; Inflammation; Cognitive Dysfunction; Dementia; Neurocognitive Disorders | interventions — Ketamine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- Ketamine (Experimental): This group received ketamine in a dose 0.5 mg / in anesthesia, in addition to other drugs used for induction, which will be standardized.
  Interventions: Drug: Ketamine
- Placebo (Placebo Comparator): This group received the equivalent volume of saline, in addition to other drugs used for induction, which will be standardized.
  Interventions: Other: Saline

INTERVENTIONS:
Drug: Ketamine
  Arms: Ketamine
Other: Saline
  Arms: Placebo

SUMMARY:
The purpose of this study is to analyze the Ketamine with its anti-inflammatory profile would be able to prevent cognitive disorders in the postoperative period of cardiac surgery, since these disorders contribute to an impact on morbidity / mortality in this population.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged over 50 years.
* Be submitted to cardiac surgery by sternotomy and with the use of cardiopulmonary bypass (CPB).
* American Society of Anesthesiologists classification 1, 2,3 and 4.

Exclusion Criteria:

* Patients undergoing reoperation.
* Patients undergoing heart transplantation.
* Patients using vasopressor agents and / or ionotropic continuous preoperatively.
* Patients with prior endotracheal intubation and consequently Ventilatory Assistance Mechanics.
* Patients with documented psychiatric disorders.
* Patients with previous cognitive disorders.
* Patients with a history of alcohol or drug abuse.
* Patients with a history of cerebrovascular accident (CVA) with less than 3 months.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-04; Primary Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Change in cognitive disorder, defined by a drop of 2 points in the Mini-Mental State Examination | Baseline and 7 days
Detectable levels of inflammatory biomarkers in bloodstream, such as: P-selectin (CD62p- ng/ml), CD40L soluble (ng/ml), s100B (ng/ml) | Change from baseline at 6 hours and 24 hours after surgery

SECONDARY OUTCOMES:
Delirium assessed using the Confusion Assessment Method (CAM) | 24 hours after surgery
Sternotomy Pain assessed using the Visual Analogue Scale | 24 hours after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Rebeca GA Andrade, master, Principal Investigator — Instituto de Medicina Integral Prof Fernando Figueira
Locations (1):
- Instituto de Medicina Integral Prof Fernando Figueira, Recife, Pernambuco, Brazil

REFERENCES:
- [Result] Hudetz JA, Iqbal Z, Gandhi SD, Patterson KM, Byrne AJ, Hudetz AG, Pagel PS, Warltier DC. Ketamine attenuates post-operative cognitive dysfunction after cardiac surgery. Acta Anaesthesiol Scand. 2009 Aug;53(7):864-72. doi: 10.1111/j.1399-6576.2009.01978.x. Epub 2009 Apr 28. PMID 19422355
- [Result] Cata JP, Abdelmalak B, Farag E. Neurological biomarkers in the perioperative period. Br J Anaesth. 2011 Dec;107(6):844-58. doi: 10.1093/bja/aer338. Epub 2011 Nov 6. PMID 22065690
- [Result] Dale O, Somogyi AA, Li Y, Sullivan T, Shavit Y. Does intraoperative ketamine attenuate inflammatory reactivity following surgery? A systematic review and meta-analysis. Anesth Analg. 2012 Oct;115(4):934-43. doi: 10.1213/ANE.0b013e3182662e30. Epub 2012 Jul 23. PMID 22826531